CLINICAL TRIAL: NCT06806761
Title: Mapping the Time Course of Recovery of Sitting and Standing Balance and Walking After Stroke
Brief Title: Tracking Balance and Walking Recovery After Stroke
Acronym: FOSTER
Status: Recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Revalidatieziekenhuis InkendaaI (Network)
Responsible Party: Principal Investigator, Eva Swinnen, Assistant Professor, Vrije Universiteit Brussel
Other Study IDs: 101136244_FOSTER
Record Dates: First submitted 2024-11-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: stroke; balance; longitudinal; gait initiation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients in the first 6 months after stroke: Participants in this study will be adults aged 18 years or older, following a supratentorial stroke, as defined by the World Health Organization (WHO). Inclusion will occur as soon as possible after hospital admission. Participants must be capable of providing informed consent, which may be written, verbal, or provided by proxy if necessary.
  Exclusion criteria include the presence of other neurological or orthopedic disorders (e.g., Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis) that impair motor function, severe complicating comorbidities imposing health risks (e.g., cardiovascular instability), significant deficits in communication, memory, or understanding (defined by a score of less than 21 on the Montreal Cognitive Assessment (MoCA)), and insufficient knowledge of Dutch, French, German, or English.
  Interventions: Other: Longitudinal prospective cohort study

INTERVENTIONS:
Other: Longitudinal prospective cohort study — Description: Patients after stroke who meet the in- and exclusion criteria will be examined up to 6 times during the first 6 months after their stroke.

SUMMARY:
This study aims to understand how balance and walking abilities recover after a stroke, using innovative tools like an interactive assessment game. By observing patients over time, the investigators seek to identify recovery patterns that can improve rehabilitation strategies tailored to individual needs.

Interacting with a game designed to assess balance and movement, participants will perform tasks involving sitting balance, standing balance, and gait initiation. The game measures aspects like reaction time, movement accuracy, and postural control, providing detailed insights into recovery progress. These data will validate prediction models to support personalized care.

The study is non-invasive, does not interfere with usual care, and prioritizes patient safety. The investigators' ultimate goal is to enhance the understanding of recovery, leading to better care and improved quality of life for stroke survivors.

DETAILED DESCRIPTION:
During this longitudinal observational study, patients following a supratentorial stroke will be included as soon as possible after admission, provided they meet the inclusion criteria. Assessments will take place at fixed time points relative to stroke onset: baseline (as soon as possible after admission) and at 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge). The study aims to investigate recovery patterns in balance and walking (gait initiation) abilities, contributing to the validation of predictive models that support personalized rehabilitation strategies.

At each time point, participants will perform standardized assessments targeting sitting balance, standing balance, and gait initiation. These assessments combine clinical scales (e.g., Fugl-Meyer Assessment for the lower limb, Berg Balance Scale, Functional Ambulation Categories) and biomechanical measurements collected using electromyography (EMG) sensors, inertial measurement units (IMUs), force plates, and a Kinect camera. EMG will provide detailed insights into muscle activation patterns, while IMUs (positioned on the sternum, pelvis, and non-paretic wrist) will measure acceleration and gyroscopic data to evaluate trunk movement and postural control. Force plates will provide data on weight distribution and stability, whereas the Kinect camera will capture posture and reaching accuracy data. An interactive assessment game will be used to evaluate task performance under various conditions, including anticipatory tasks (where the target location is known), reactive tasks (requiring quick adjustments to unpredictable targets), and cognitive-motor dual-task scenarios (involving decision-making under time pressure). Data from these assessments will provide detailed insights into recovery processes.

In addition to in-lab assessments, the study will also evaluate the relationship between laboratory-based measures and real-world functional activity. Participants will wear an activity monitor for three days following the longitudinal assessment sessions to measure real-world activity, including time spent sitting, standing, and walking. This approach allows the investigators to explore how improvements observed in the lab translate into functional recovery in daily life.

By combining clinical, biomechanical, and real-world data, the study seeks to address gaps in stroke recovery research, particularly the factors influencing recovery trajectories and how rehabilitation can be optimized. The findings are expected to enhance understanding of recovery patterns, inform individualized rehabilitation plans, and ultimately improve quality of life for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Diagnosis of supratentorial stroke (as defined by the WHO)
* Able to provide written or verbal informed consent (written, verbal or by proxy)

Exclusion Criteria:

* Other neurological/orthopedic disorders (e.g., Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis) leading to impairments in motor function.
* Severe complicating comorbidities imposing health risks (e.g., cardiovascular instability)
* Severe deficits in communication, memory or understanding (Montreal Cognitive Assessment test (MoCA) < 21); and
* Insufficient knowledge of Dutch, French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the first 6 months after stroke: Participants in this study will be adults aged 18 years or older, following a supratentorial stroke, as defined by the World Health Organization (WHO).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2028-12-09 (Estimated); Study Completion 2028-12-09 (Estimated)

PRIMARY OUTCOMES:
Postural control | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Postural control during dynamic tasks (sitting, standing, gait initiation) measured using wearable sensors (e.g., IMUs) and other biomechanical measurement systems (e.g., force plates, Kinect cameras).
Weight distribution | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Weight distribution during balance and movement tasks (standing, gait initiation) using force plates.
Movement coordination | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Movement coordination assessed during functional motor tasks (sitting, standing, gait initiation) using wearable sensors (e.g., IMUs), force plates, and Kinect camera.
Neuromuscular activity | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Neuromuscular activity evaluated during dynamic tasks (sitting, standing, gait initiation) using muscle activity measurement systems (e.g., EMG sensors).

SECONDARY OUTCOMES:
Reaction time | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Time from target appearance to reaching/stepping movement initiation during sitting balance, standing balance, and gait initiation tasks, measured using the interactive assessment game and Kinect camera.
Movement time | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Duration of the reaching/stepping movement from initiation to completion during sitting balance, standing balance, and gait initiation tasks, measured using the interactive assessment game and Kinect camera.
Reaching or stepping accuracy | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Number of successful target reaches during sitting and standing balance tasks, and correct leg usage during gait initiation tasks, measured using the Kinect camera and the interactive assessment game.
Upper limb dynamics | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Acceleration of upper limb movements during sitting and standing reaching tasks, measured using an IMU sensor on the wrist.
Error rate during dual-task performance | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Frequency of incorrect responses during Go/No-Go tasks integrated into sitting and standing tasks, measured using the interactive assessment game and Kinect camera.
Daily activity monitoring | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Measurement of time spent sitting, standing, and walking using the Activ8 sensor over a continuous 3-day monitoring period after each assessment.
Lower limb motor impairment | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Fugl-Meyer Assessment of the lower limb (FMA LL). Scores ranging from 0 to 34 (no motor impairment present).
Lower limb strength | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Motricity Index of the lower limb (MI LL). Scores ranging from 0 (no movement) to 99 (normal power).
Dynamic sitting balance | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Trunk Impairment Scale (TIS), items D.1 till D.6. Scores ranging from 0 to 6 (no balance impairment present).
Dynamic standing balance | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  The Mini-BESTest and/or the Berg Balance Scale (BBS), depending on the Functional Ambulation Categories (FAC)-score. Scores ranging from 0 (severe balance deficits) to 28 (normal balance) and/or from 0 (severe balance deficits) to 56 (normal balance), respectively.
Walking independence | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Functional Ambulation Categories (FAC)-score, ranging from 0 (not able to walk) to 5 (independent ambulator who can walk freely on any surface).
Walking performance | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  10-meter walk test (10MWT), measuring the comfortable and maximum walking speed over a 10 meter walking distance.
Daily life functioning | Baseline
  Modified Ranking Scale (mRS), both premorbid (pre-stroke) and baseline (post-stroke). Scores ranging from 0 (no symptoms) to 5 (severe disability).
Activities of daily living | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Functional Independence Measure (FIM), ranging from 18 (complete dependence/total assistance) to 126 (complete independence).
Cognitive functioning | Baseline (screening)
  Montreal Cognitive Assessment (MoCA), ranging from 0 to 30. A score lower than or equal to 21 is suggesting that the patient is not able to take part in our study.
Mental health | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  Hospital Anxiety and Depression Scale (HADS), with separate scores for anxiety and depression. Both subscale scores are ranging from 0 to 21. A total score is calculated by adding together all the values, with a total score ≥ 12 suggesting depression, whereas sub-scores of ≥ 8 suggest anxiety or depression.
Health-related quality of life | Baseline, 3, 5, 8, 12, and 24 weeks post-stroke (or until discharge)
  36-item Short Form survey (SF-36), ranging from 0 to 100, with higher scores defining a more favorable health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Inkendaal rehabilitation hospital, Sint-Pieters-Leeuw, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
This study is part of the EU Horizon 2020 TARGET project, following its DMP to ensure data is handled ethically, legally, and sustainably in line with FAIR principles (Findability, Accessibility, Interoperability, Reusability). The plan ensures systematic organization, quality consistency via standardized procedures, and compliance with GDPR, national laws, and EU requirements. Personal data is processed securely, only when necessary for project objectives, with approvals and written consent from participants. Methods include interviews, surveys, workshops, and questionnaires. Data is stored with robust backup and preservation strategies to prevent loss and ensure future usability. Sharing is (currently) restricted to the consortium under a signed data transfer agreement, with external sharing undecided. Data not publicly available includes: third-party data without permission for public release, data compromising IP protection, and participant data that cannot be fully anonymized.
Supporting Information: Study Protocol, SAP, CSR